CLINICAL TRIAL: NCT03041025
Title: A Multi-center, Randomized, Double-blind (Sponsor Open), Placebo-controlled, Repeat-dose, Proof of Mechanism Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Explore Efficacy of GSK2330811 in Participants With Diffuse Cutaneous Systemic Sclerosis
Brief Title: Proof of Mechanism Study of GSK2330811 in Diffuse Cutaneous Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201247; 2016-003417-95 (EudraCT Number)
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Scleroderma, Systemic
Keywords: Systemic Sclerosis; Repeat-dose; Phase IIA; GSK2330811; Pharmacodynamics; Pharmacokinetics; Proof of mechanism study
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: GSK2330811 100 mg (Experimental): During Cohort 1, participants will receive a single dose of GSK2330811 100 mg by SC injection via needle and syringe in to the abdomen, thigh or upper arm by the investigator or designee at every other week from D1 to D71 (total 6 doses) for 10 weeks. Participants will be followed-up up to W28 D197.
  Interventions: Drug: GSK2330811
- Cohort 2: GSK2330811 300 mg (Experimental): During Cohort 2, participants will receive a single dose of GSK2330811 300 mg by SC injection (3 vials of 1 mL each of GSK2330811 100 mg) via needle and syringe in to the abdomen, thigh or upper arm by the investigator or designee at every other week from D1 to D71 (total 6 doses) for 10 weeks. Participants will be followed-up up to W28 D197.
  Interventions: Drug: GSK2330811
- Cohort 1: Placebo (Placebo Comparator): During Cohort 1, participants will receive a single dose of placebo by SC injection via needle and syringe in to the abdomen, thigh or upper arm by the investigator or designee at every other week from D1 to D71 (total 6 doses) for 10 weeks. Participants will be followed-up up to W28 D197.
  Interventions: Drug: Placebo
- Cohort 2: Placebo (Placebo Comparator): During Cohort 2, participants will receive a single dose of placebo by SC injection (3 vials of 1 mL each) via needle and syringe in to the abdomen, thigh or upper arm by the investigator or designee at every other week from D1 to D71 (total 6 doses) for 10 weeks. Participants will be followed-up up to W28 D197.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2330811 — GSK2330811 will be provided in vials and packed in 1 vial per carton. Each vial will contain 1.2 mL fill with 1 mL extractable volume at 100 mg/mL.
  Arms: Cohort 1: GSK2330811 100 mg; Cohort 2: GSK2330811 300 mg
Drug: Placebo — Normal saline (0.9 percent weight per volume sodium chloride).
  Arms: Cohort 1: Placebo; Cohort 2: Placebo

SUMMARY:
GSK2330811 is a humanized monoclonal antibody which is in development for systemic sclerosis (SSc), a rare autoimmune disease with high morbidity and mortality. Currently, there are no approved disease modifying therapies and it is an area of high unmet medical need. GSK2330811 has been shown to bind and neutralize Oncostatin M (OSM) that has been associated with fibrosis, vasculopathy and inflammation in a number of diseases. This multi-center, randomized, double-blind (sponsor open), placebo controlled, proof of mechanism study will be the first study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of repeat subcutaneous (SC) doses of GSK2330811 in male and female participants with diffuse cutaneous SSc (dcSSc). Participants with active disease and a disease duration of <= 60 months will be enrolled. Approximately 24 to 40 participants will be randomized across two sequential cohorts. Cohort 1 will evaluate a repeat-dose predicted to provide sub-maximal inhibition of OSM, leading to a dose escalation decision. Cohort 1 is planned to consist of at least 4 participants, randomized such that 3 participants will receive GSK2330811 100 milligram (mg) and 1 will receive placebo. Cohort 2 is planned to consist of at least 20 participants, randomized such that participants will receive GSK2330811 300 mg and placebo in a 3:1 ratio respectively. The duration of the study is up to 34 weeks including a screening period of up to 6 weeks, treatment period of 12 weeks and follow-up period of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants of 18 years or over, at the time of signing the informed consent.
* Documented diagnosis of systemic sclerosis with diffuse cutaneous involvement.
* Modified rodnan skin score (mRSS) >=10 and <=35 at screening.
* In all cases, a disease duration of <=60 months at screening, defined as time from onset of the first non-Raynaud's phenomenon manifestation.
* Active disease defined by at least one of the following criteria at screening:

  * C-Reactive Protein (CRP) >=6 mg/liter (L) (0.6 mg/deciliter [dL]), that in the opinion of the investigator is due to SSc.
  * Disease duration <=18 months at screening, defined as time from the first non-Raynaud's phenomenon manifestation.
  * Increase of >=3 mRSS units, compared with an assessment performed within the previous 6 months.
  * Involvement of one new body area and an increase of >=2 mRSS units compared with an assessment performed within the previous 6 months.
  * Involvement of two new body areas within the previous 6 months.
* An area of uninvolved or mildly thickened skin that in the opinion of the investigator would allow subcutaneous injection either at abdomen, front or middle region of the thigh or at outer area of the upper arm.
* An area of involved skin (mRSS >=1) on the forearm suitable for repeated skin biopsies to be collected.
* Participants who are taking mycophenolate mofetil (<=3,000 mg/day) or equivalent mycophenolate sodium (<=2160 mg/day) are permitted in the study if the participant has been on a stable dose for >=3 months at the first dosing day (Day 1) and participant and investigator are willing to continue this dose until at least completion of the Day 85 (Week 12) visit. If mycophenolate was recently ceased, there must be >=3 months between the date mycophenolate was ceased and the first dosing day (Day 1).
* Participants who are taking oral corticosteroids (<=10 mg/day of prednisone or equivalent) are permitted in the study if the participant has been receiving a dose no greater than 10 mg/day for at least 4 weeks at the first dosing day (Day 1) and the investigator does not anticipate increasing the dose above 10 mg/day during the study.
* Participants who are taking phosphodiesterase 5 (PDE5) inhibitors and endothelin receptor antagonists (including bosentan) are permitted in the study if the participant has been on a stable dose for at least 4 weeks for PDE5 inhibitors and for at least 3 months for endothelin antagonists at the first dosing day (Day 1) and participant and investigator are willing to continue this dose until at least completion of the Day 85 (Week 12) visit.
* Participants who are taking non-immunosuppressive medications are permitted in the study (e.g. hydroxychloroquine, angiotensin converting enzyme (ACE) inhibitors/angiotensin II receptor (AR) blockers, calcium-channel blockers and proton-pump inhibitors). However no new long-term medications and no dose-changes to existing long term medications are permitted during the two weeks prior to the first dosing day (Day 1).
* Male participants must agree to use contraception during the dosing period and for at least 126 days (18 weeks) after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and either she is not a woman of childbearing potential (WOCBP) or she is a WOCBP who agrees to use contraceptives from 28 days prior to first dosing day (Day 1), during the dosing period and for at least 126 days (18 weeks) after the last dose of study treatment.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions for this study.

Exclusion Criteria:

* Participants classified to the limited cutaneous SSc subset, as determined by the investigator.
* Rheumatic autoimmune disease other than dcSSc including but not limited to rheumatoid arthritis, systemic lupus erythematosus, mixed connective tissue disorder, polymyositis, dermatomyositis, systemic vasculitis and primary Sjogren's syndrome, as determined by the investigator.
* Forced vital capacity (FVC) <=50 percentage of predicted, or a diffusing capacity of the lung for carbon dioxide (DLCO) (corrected for hemoglobin) <=40 percentage of predicted at screening.
* Pulmonary arterial hypertension, as determined by the investigator.
* Clinically significant inflammatory myositis (related to SSc), as determined by the investigator.
* SSc renal crisis within 6 months of the first day of dosing (Day 1).
* History of clinically significant or uncontrolled cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease at screening not related to SSc and that in the opinion of the investigator would prevent participation in the study.
* Known bleeding or coagulation disorder.
* Major surgery (including joint surgery) within 3 months prior to screening, or planned during the duration of the study.
* Clinically significant multiple or severe drug allergies (including to humanized monoclonal antibodies), intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* An active infection, or a history of infections as follows:

  * History of opportunistic infections that have not resolved by 6 months prior to the first day of dosing (Day1) or recurrent infection as determined by the investigator. This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless it is of an unusual severity or frequency.
  * A serious infection requiring treatment with intravenous antibiotics and/or hospitalization, if the last dose of antibiotics or the hospital discharge date was within 3 months of the first day of dosing (Day1).
  * An acute or chronic infection requiring treatment with oral antibiotics or antiviral medications, if the last dose was received within 4 weeks of the first day of dosing (Day1).
  * Any active or unresolved bacterial, viral or fungal infection present on the first day of dosing (Day1), whether requiring treatment or not. This does not include fungal nail infections.
  * Active or past osteomyelitis, unless fully resolved in the opinion of the investigator.
  * Symptomatic herpes zoster that has not resolved by 3 months prior to the first day of dosing (Day1).
  * History of Tuberculosis (TB) or a positive QuantiFERON-TB Gold test or QuantiFERON-TB Gold PLUS test at screening.
* If the QuantiFERON-TB Gold test or QuantiFERON-TB Gold PLUS test is indeterminate, it can be repeated once. A participant will not be eligible unless the second test is negative or they have a negative tuberculin skin test (defined as skin induration <5 mm at 48 to 72 hours, regardless of Bacillus Calmette-Guerin or other vaccination history).
* There must be no other clinical evidence of TB on physical examination of the participant (screening examination).
* Alanine transferase (ALT) >2 times upper limit of normal (ULN) at screening.
* Bilirubin >1.5 times ULN at screening (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percentage).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of gilbert's syndrome or asymptomatic gallstones). Participants with evidence of liver fat on imaging but who are otherwise eligible for the study criteria may be enrolled.
* QTc >480 milliseconds (msec) or QTc >500 msec in participants with bundle branch block at screening.
* A history of carcinoma in situ and malignant disease, with the exception of basal cell carcinoma that has been completely excised prior to the study.
* Treatment with methotrexate within 3 months prior to the first dosing day (Day 1).
* Previous or planned bone marrow transplant (e.g. autologous stem cell transplant).
* Treatment with a biologic within the following timeframes:

  * Tocilizumab, abatacept or anti- tumor necrosis factor (including etanercept, infliximab, certolizumab, golimumab or adalimumab) within 3 months prior to the first dosing day (Day 1).
  * Rituximab within 12 months prior to the first dosing day (Day 1).
  * For any other biologic consult the medical monitor.
* Treatment with oral or intravenous cyclophosphamide within 6 months prior to the first dosing day (Day 1).
* Treatment with any other non-biologic systemic immunosuppressive medication (e.g. azathioprine, tacrolimus, ciclosporin) not mentioned above within 4 weeks prior to the first dosing day (Day 1), with the exception of mycophenolate and permitted oral corticosteroid.
* Treatment with topical immunosuppressive medications (e.g. topical corticosteroids, tacrolimus) within 1 week prior to the first dosing day (Day 1).
* Treatment with intravenous prostanoids (e.g. iloprost) within 2 weeks prior to the first dosing day (Day 1) or planned treatment before the Day 85 (Week 12) visit.
* Treatment with anti-fibrotic medications including tyrosine kinase inhibitors (e.g. nintedinib and imatinib) and pirfenidone within 3 months prior to the first dosing day (Day 1).
* Live vaccine(s) within 4 weeks prior to the first dosing day (Day 1), or plans to receive such vaccines during the study.
* Treatment with anti-coagulant medications, including warfarin, heparin, thrombin inhibitors, and factor Xa inhibitors within 2 weeks prior to the first dosing day (Day 1).
* Treatment with anti-platelet medications (e.g. clopidogrel, prasugrel, ticagrelor and dipyridamole) within 2 weeks prior to first dosing day (Day 1). This does not include aspirin at doses of 150 mg or less, or non-steroidal anti-inflammatory drugs, which are permitted.
* Current enrollment or past participation within the last 30 days before signing of consent in any other clinical study involving an investigational study treatment.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day (Day 1).
* Any of the following at screening:

  * Hemoglobin <110 gram (g)/L
  * Platelet count <150x10^9/L
  * Estimated glomerular filtration rate (GFR) (modification of diet in renal disease [MDRD] calculation) of <45 mL/minute/1.73m^2
* A positive human immunodeficiency virus (HIV) antibody test at screening.
* Presence of hepatitis B surface antigen (HBsAg) at screening.
* Positive hepatitis B core antibody (HBcAb) test at screening.
* Positive hepatitis C antibody test result at screening or within 3 months prior to starting study treatment.
* Positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Sensitivity to any of the study treatments or components thereof, or other allergy that in the opinion of the investigator, contraindicates participation in the study.
* Where participation in the study would result in donation of blood or blood products in excess of a volume of 500 mL during the study.
* A history of drug and alcohol misuse that could interfere with participation in the trial according to the protocol, or in the opinion of the investigator impacts on the physical or mental wellbeing of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (6):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
- GSK Investigational Site, Toronto, Ontario, Canada
- GSK Investigational Site, Nijmegen, Netherlands
- United Kingdom (6):
  - GSK Investigational Site, Salford, Greater Manchester
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Denton CP, Del Galdo F, Khanna D, Vonk MC, Chung L, Johnson SR, Varga J, Furst DE, Temple J, Zecchin C, Csomor E, Lee A, Wisniacki N, Flint SM, Reid J. Biological and clinical insights from a randomized phase 2 study of an anti-oncostatin M monoclonal antibody in systemic sclerosis. Rheumatology (Oxford). 2022 Dec 23;62(1):234-242. doi: 10.1093/rheumatology/keac300. PMID 35583273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind (sponsor open), proof of mechanism study of GSK2330811 in participants with diffuse cutaneous systemic sclerosis. This study was conducted in Canada, Netherlands, United Kingdom and United States.
Pre-assignment Details: A total of 35 participants were enrolled in this study.
Groups:
- Placebo: Participants received subcutaneous injection of placebo on Day 1 and then every other week until the final dose on Day 71 (Week 10).
- GSK2330811 100 mg: Participants received subcutaneous injection of GSK2330811 100 milligrams (mg) on Day 1 and then every other week until the final dose on Day 71 (Week 10).
- GSK2330811 300 mg: Participants received subcutaneous injection of GSK2330811 300 mg on Day 1 and then every other week until the final dose on Day 71 (Week 10).
Period: Overall Study
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Started | 8 | 3 | 24
Completed | 7 | 3 | 22
Not Completed | 1 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg | Total
Number analyzed (Participants) | 8 | 3 | 24 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (15.42) | 66.7 (4.73) | 52.6 (12.59) | 53.4 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 19 | 26
  Male | 2 | 2 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 1 | 1
  Asian - East Asian Heritage | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 3 | 3
  White - White/Caucasian/European Heritage | 7 | 3 | 20 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician. SAEs were collected up to Day 197, but the protocol also allowed investigators to report SAEs occurring after participants had completed the study. This outcome measure includes two SAEs reported after participants had completed the study, occurring on Day 306 and Day 603 following first dose. Safety Population consisted of all randomized participants who have taken at least 1 dose of study treatment.
Time Frame: Up to Day 197, but protocol allowed for additional events to be collected; up to Day 603 post first dose
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 24
Participants
  Non-SAEs | 8 | 3 | 24
  SAEs | 1 | 0 | 2

2. Primary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count, White Blood Cell (WBC) Count
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, Platelet Count and WBC count. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Giga cells per liter
  Day 15: Basophils, n=8,3,23 | -0.006 (0.0262) | 0.013 (0.0252) | 0.007 (0.0325)
  Day 29: Basophils, n=8,3,23 | -0.005 (0.0288) | -0.003 (0.0252) | 0.003 (0.0350)
  Day 43: Basophils, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Basophils, n=8,3,22 | -0.005 (0.0169) | 0.027 (0.0635) | -0.005 (0.0323)
  Day 57: Basophils, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Basophils, n=6,3,22 | -0.010 (0.0167) | 0.013 (0.0404) | -0.004 (0.0333)
  Day 71: Basophils, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: Basophils, n=8,3,20 | -0.010 (0.0267) | -0.003 (0.0208) | -0.008 (0.0341)
  Day 85: Basophils, n=7,2,22: number analyzed (Participants) | 7 | 2 | 22
  Day 85: Basophils, n=7,2,22 | -0.020 (0.0294) | 0.045 (0.0636) | 0.000 (0.0344)
  Day 113: Basophils, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 113: Basophils, n=7,3,21 | -0.006 (0.0237) | 0.040 (0.0693) | -0.002 (0.0390)
  Day 155: Basophils, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: Basophils, n=7,3,20 | 0.004 (0.0270) | 0.060 (0.0721) | 0.000 (0.0400)
  Day 197: Basophils, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 197: Basophils, n=7,3,18 | -0.006 (0.0399) | 0.033 (0.0208) | 0.015 (0.0517)
  Day 15: Eosinophils, n=8,3,23 | 0.016 (0.0616) | 0.070 (0.0700) | 0.084 (0.2934)
  Day 29: Eosinophils, n=8,3,23 | 0.036 (0.0901) | 0.060 (0.2007) | 0.001 (0.1633)
  Day 43: Eosinophils, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Eosinophils, n=8,3,22 | 0.019 (0.0500) | 0.103 (0.1026) | -0.015 (0.1954)
  Day 57: Eosinophils, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Eosinophils, n=6,3,22 | 0.010 (0.0473) | 0.113 (0.1795) | -0.034 (0.1797)
  Day 71: Eosinophils, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: Eosinophils, n=8,3,20 | 0.018 (0.0440) | 0.137 (0.2344) | 0.012 (0.1241)
  Day 85: Eosinophils, n=7,2,22: number analyzed (Participants) | 7 | 2 | 22
  Day 85: Eosinophils, n=7,2,22 | 0.001 (0.0406) | 0.130 (0.3111) | -0.035 (0.1773)
  Day 113: Eosinophils, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 113: Eosinophils, n=7,3,21 | 0.056 (0.1005) | 0.070 (0.0872) | 0.087 (0.2873)
  Day 155: Eosinophils, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: Eosinophils, n=7,3,20 | 0.003 (0.0403) | 0.080 (0.0300) | 0.005 (0.1695)
  Day 197: Eosinophils, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 197: Eosinophils, n=7,3,18 | 0.069 (0.1426) | 0.170 (0.1323) | 0.056 (0.1302)
  Day 15: Lymphocytes, n=8,3,23 | -0.116 (0.3926) | 0.103 (0.3955) | -0.125 (0.4110)
  Day 29: Lymphocytes, n=8,3,23 | -0.064 (0.2539) | 0.477 (0.4177) | -0.102 (0.6071)
  Day 43: Lymphocytes, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Lymphocytes, n=8,3,22 | 0.020 (0.2891) | 0.530 (0.3270) | -0.078 (0.6156)
  Day 57: Lymphocytes, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Lymphocytes, n=6,3,22 | -0.043 (0.3732) | 0.563 (0.3798) | 0.105 (0.5853)
  Day 71: Lymphocytes, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: Lymphocytes, n=8,3,20 | -0.060 (0.2384) | 0.430 (0.3601) | 0.155 (0.5169)
  Day 85: Lymphocytes, n=7,2,22: number analyzed (Participants) | 7 | 2 | 22
  Day 85: Lymphocytes, n=7,2,22 | -0.109 (0.2202) | 0.580 (0.4667) | 0.313 (0.5521)
  Day 113: Lymphocytes, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 113: Lymphocytes, n=7,3,21 | -0.297 (0.5087) | 0.383 (0.3907) | 0.287 (0.6783)
  Day 155: Lymphocytes, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: Lymphocytes, n=7,3,20 | -0.046 (0.2327) | 0.160 (0.2600) | 0.202 (0.4504)
  Day 197: Lymphocytes, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 197: Lymphocytes, n=7,3,18 | -0.066 (0.4108) | -0.010 (0.4419) | 0.039 (0.7780)
  Day 15: Monocytes, n=8,3,23 | 0.096 (0.1507) | -0.017 (0.1102) | -0.051 (0.1659)
  Day 29: Monocytes, n=8,3,23 | 0.006 (0.0578) | -0.030 (0.3959) | -0.120 (0.2175)
  Day 43: Monocytes, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Monocytes, n=8,3,22 | 0.103 (0.2093) | 0.047 (0.1069) | -0.106 (0.2045)
  Day 57: Monocytes, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Monocytes, n=6,3,22 | -0.037 (0.0698) | -0.120 (0.1600) | -0.130 (0.2216)
  Day 71: Monocytes, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: Monocytes, n=8,3,20 | 0.050 (0.1414) | -0.003 (0.0404) | -0.070 (0.1838)
  Day 85: Monocytes, n=7,2,22: number analyzed (Participants) | 7 | 2 | 22
  Day 85: Monocytes, n=7,2,22 | -0.007 (0.0652) | 0.140 (0.1697) | -0.127 (0.2495)
  Day 113: Monocytes, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 113: Monocytes, n=7,3,21 | 0.070 (0.1494) | 0.030 (0.1735) | -0.028 (0.2246)
  Day 155: Monocytes, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: Monocytes, n=7,3,20 | 0.064 (0.1229) | 0.167 (0.1250) | -0.022 (0.1414)
  Day 197: Monocytes, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 197: Monocytes, n=7,3,18 | 0.051 (0.2242) | -0.043 (0.1266) | -0.053 (0.2234)
  Day 15: Total neutrophils, n=8,3,23 | 0.228 (1.3240) | 1.060 (3.0143) | -0.917 (1.4114)
  Day 29: Total neutrophils, n=8,3,23 | 0.318 (1.4309) | 0.323 (1.8591) | -1.104 (1.4251)
  Day 43: Total neutrophils, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Total neutrophils, n=8,3,22 | 0.315 (1.3403) | -0.350 (1.4731) | -1.406 (1.4631)
  Day 57: Total neutrophils, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Total neutrophils, n=6,3,22 | 0.538 (0.9156) | -0.517 (1.9998) | -1.387 (1.4428)
  Day 71: Total neutrophils, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: Total neutrophils, n=8,3,20 | 0.789 (2.1739) | -0.223 (1.8928) | -1.369 (1.6361)
  Day 85: Total neutrophils, n=7,2,22: number analyzed (Participants) | 7 | 2 | 22
  Day 85: Total neutrophils, n=7,2,22 | -0.139 (1.1995) | -0.990 (2.9698) | -1.424 (2.3949)
  Day 113: Total neutrophils, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: Total neutrophils, n=7,3,20 | 0.680 (1.2472) | -0.263 (1.0384) | -1.002 (1.5195)
  Day 155: Total neutrophils, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: Total neutrophils, n=7,3,20 | 0.027 (1.2229) | -0.673 (2.1324) | -0.183 (1.2208)
  Day 197: Total neutrophils, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 197: Total neutrophils, n=7,3,18 | 0.317 (1.3578) | -1.603 (4.0868) | -0.001 (1.4937)
  Day 15: Platelet count, n=8,3,23 | -1.5 (24.02) | -42.0 (32.70) | -124.6 (87.57)
  Day 29: Platelet count, n=7,3,23: number analyzed (Participants) | 7 | 3 | 23
  Day 29: Platelet count, n=7,3,23 | -5.9 (20.38) | -39.7 (29.28) | -145.7 (94.01)
  Day 43: Platelet count, n=8,3,23 | -16.1 (14.56) | -49.0 (22.27) | -150.2 (90.41)
  Day 57: Platelet count, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Platelet count, n=6,3,22 | -4.2 (20.40) | -66.0 (42.04) | -148.6 (90.99)
  Day 71: Platelet count, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 71: Platelet count, n=7,3,20 | -12.3 (17.67) | -41.7 (45.21) | -129.4 (90.54)
  Day 85: Platelet count, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: Platelet count, n=7,3,22 | -18.0 (25.89) | -48.0 (29.10) | -97.4 (73.99)
  Day 113: Platelet count, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: Platelet count, n=7,3,20 | -14.4 (25.53) | -20.3 (42.52) | -61.2 (96.89)
  Day 155: Platelet count, n=6,3,20: number analyzed (Participants) | 6 | 3 | 20
  Day 155: Platelet count, n=6,3,20 | -26.7 (19.62) | 15.0 (31.24) | -6.9 (60.00)
  Day 197: Platelet count, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: Platelet count, n=7,3,19 | -10.1 (30.30) | -20.7 (71.53) | -10.3 (42.86)
  Day 15: WBC count, n=8,3,23 | 0.20 (1.546) | 1.20 (2.685) | -1.00 (1.487)
  Day 29: WBC count, n=8,3,23 | 0.28 (1.400) | 0.80 (1.212) | -1.33 (1.927)
  Day 43: WBC count, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: WBC count, n=8,3,22 | 0.46 (1.418) | 0.33 (0.950) | -1.60 (2.039)
  Day 57: WBC count, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: WBC count, n=6,3,22 | 0.43 (0.774) | 0.03 (1.617) | -1.46 (1.947)
  Day 71: WBC count, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: WBC count, n=8,3,20 | 0.76 (2.191) | 0.33 (1.258) | -1.29 (1.953)
  Day 85: WBC count, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: WBC count, n=7,3,22 | -0.29 (1.182) | -0.10 (1.400) | -1.27 (2.509)
  Day 113: WBC count, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 113: WBC count, n=7,3,21 | 0.47 (1.138) | 0.27 (0.473) | -0.61 (1.913)
  Day 155: WBC count, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: WBC count, n=7,3,20 | 0.07 (1.228) | -0.20 (1.778) | 0.01 (1.571)
  Day 197: WBC count, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: WBC count, n=7,3,19 | 0.31 (1.469) | -1.50 (4.444) | -0.01 (1.948)

3. Primary Outcome: Change From Baseline in Hematology Parameters: Hemoglobin, Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Blood samples were collected to analyze the hematology parameters: hemoglobin and MCHC. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Grams per liter
  Day 15: Hemoglobin, n=8,3,23 | -2.8 (8.89) | 2.0 (7.00) | -0.2 (5.31)
  Day 29: Hemoglobin, n=8,3,23 | -2.5 (6.55) | -0.7 (11.06) | -3.7 (7.45)
  Day 43: Hemoglobin, n=8,3,23 | -2.5 (6.39) | -1.7 (8.50) | -7.7 (9.06)
  Day 57: Hemoglobin, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Hemoglobin, n=6,3,22 | -3.8 (8.47) | -2.7 (11.15) | -13.7 (12.32)
  Day 71: Hemoglobin, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: Hemoglobin, n=8,3,20 | -4.1 (10.38) | -6.3 (4.73) | -21.2 (11.61)
  Day 85: Hemoglobin, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: Hemoglobin, n=7,3,22 | -3.9 (7.58) | -10.7 (6.11) | -22.0 (10.05)
  Day 113: Hemoglobin, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 113: Hemoglobin, n=7,3,21 | -5.0 (8.43) | -9.0 (7.55) | -21.3 (10.49)
  Day 155: Hemoglobin, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: Hemoglobin, n=7,3,20 | -6.3 (9.41) | -7.3 (6.03) | -14.3 (8.62)
  Day 197: Hemoglobin, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: Hemoglobin, n=7,3,19 | -4.1 (8.88) | -6.7 (2.08) | -5.8 (6.58)
  Day 15: MCHC, n=8,3,23 | 0.9 (8.53) | -5.0 (3.00) | 2.4 (7.83)
  Day 29: MCHC, n=8,3,23 | -3.6 (6.39) | 2.0 (13.11) | 2.0 (8.30)
  Day 43: MCHC, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: MCHC, n=8,3,22 | -1.3 (9.27) | 1.0 (7.55) | 2.5 (4.86)
  Day 57: MCHC, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: MCHC, n=6,3,22 | -1.2 (10.11) | 3.7 (4.93) | 2.8 (8.42)
  Day 71: MCHC, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: MCHC, n=8,3,20 | 2.3 (12.87) | 2.7 (6.81) | 0.5 (8.62)
  Day 85: MCHC, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: MCHC, n=7,3,22 | 3.3 (10.53) | -1.7 (9.50) | 2.8 (6.68)
  Day 113: MCHC, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: MCHC, n=7,3,20 | -0.4 (7.18) | 5.0 (8.19) | -3.3 (8.16)
  Day 155: MCHC, n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: MCHC, n=7,3,17 | -1.4 (5.26) | 3.7 (4.16) | -4.2 (9.35)
  Day 197: MCHC, n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: MCHC, n=7,3,15 | -0.4 (8.58) | -0.3 (7.02) | -3.5 (8.18)

4. Primary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Proportion of red blood cells in blood
  Day 15: n=8,3,23 | -0.0089 (0.02744) | 0.0127 (0.02203) | -0.0035 (0.01771)
  Day 29: n=8,3,23 | -0.0023 (0.01955) | -0.0027 (0.04234) | -0.0141 (0.02486)
  Day 43: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: n=8,3,22 | -0.0049 (0.01788) | -0.0057 (0.03564) | -0.0271 (0.03187)
  Day 57: n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: n=6,3,22 | -0.0092 (0.02500) | -0.0120 (0.03274) | -0.0444 (0.04224)
  Day 71: n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: n=8,3,20 | -0.0146 (0.02870) | -0.0217 (0.02329) | -0.0637 (0.03983)
  Day 85: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: n=7,3,22 | -0.0151 (0.02591) | -0.0300 (0.01803) | -0.0688 (0.03265)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | -0.0141 (0.03007) | -0.0323 (0.02822) | -0.0602 (0.02839)
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | -0.0164 (0.03169) | -0.0263 (0.01626) | -0.0349 (0.02482)
  Day 197: n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: n=7,3,15 | -0.0111 (0.02634) | -0.0193 (0.00981) | -0.0125 (0.02252)

5. Primary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin (MCH)
Description: Blood samples were collected to analyze the hematology parameter: MCH. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Picogram
  Day 15: n=8,3,23 | -0.08 (0.711) | 0.03 (0.493) | 0.04 (0.503)
  Day 29: n=8,3,23 | -0.24 (0.616) | 0.37 (0.709) | -0.23 (0.437)
  Day 43: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: n=8,3,22 | -0.23 (0.807) | -0.10 (0.173) | -0.41 (0.450)
  Day 57: n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: n=6,3,22 | -0.25 (0.750) | 0.10 (0.361) | -0.39 (0.493)
  Day 71: n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: n=8,3,20 | 0.18 (0.945) | 0.17 (0.379) | -0.50 (0.503)
  Day 85: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: n=7,3,22 | 0.07 (1.034) | -0.30 (0.755) | -0.45 (0.709)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | -0.06 (0.808) | 0.87 (0.513) | -0.27 (0.873)
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | -0.16 (0.637) | 0.90 (0.200) | 0.04 (1.180)
  Day 197: n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: n=7,3,15 | -0.44 (1.015) | 0.33 (0.208) | -0.23 (1.285)

6. Primary Outcome: Change From Baseline in Hematology Parameters: Mean Corpuscle Volume (MCV), Mean Platelet Volume (MPV)
Description: Blood samples were collected to analyze the hematology parameters: MCV and MPV. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Femtoliter
  Day 15: MCV, n=8,3,23 | -0.63 (1.188) | 1.33 (1.528) | -0.39 (1.725)
  Day 29: MCV, n=8,3,23 | 0.38 (1.188) | 0.33 (1.155) | -1.17 (2.188)
  Day 43: MCV, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: MCV, n=8,3,22 | -0.38 (2.326) | -0.67 (1.528) | -1.86 (1.583)
  Day 57: MCV, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: MCV, n=6,3,22 | -0.17 (2.787) | -1.00 (0.000) | -1.77 (2.308)
  Day 71: MCV, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: MCV, n=8,3,20 | -0.13 (3.441) | -0.67 (1.528) | -1.60 (2.722)
  Day 85: MCV, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: MCV, n=7,3,22 | -0.71 (1.113) | -0.67 (0.577) | -2.05 (2.478)
  Day 113: MCV, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 113: MCV, n=7,3,21 | -0.29 (2.563) | 1.00 (1.732) | 0.00 (3.225)
  Day 155: MCV, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: MCV, n=7,3,20 | -0.14 (1.215) | 1.67 (0.577) | 1.26 (4.584)
  Day 197: MCV, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 197: MCV, n=7,3,18 | -1.29 (1.799) | 0.67 (2.082) | -0.02 (3.575)
  Day 15: MPV, n=8,3,23 | 0.04 (0.256) | 0.20 (0.361) | 0.45 (0.460)
  Day 29: MPV, n=8,3,23 | -0.04 (0.378) | 0.47 (0.764) | 0.29 (0.630)
  Day 43: MPV, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 43: MPV, n=7,3,22 | -0.14 (0.276) | 0.23 (0.737) | 0.07 (0.594)
  Day 57: MPV, n=6,3,21: number analyzed (Participants) | 6 | 3 | 21
  Day 57: MPV, n=6,3,21 | 0.23 (0.446) | 0.47 (0.416) | 0.12 (0.599)
  Day 71: MPV, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 71: MPV, n=7,3,20 | -0.21 (0.393) | 0.23 (0.231) | -0.15 (0.516)
  Day 85: MPV, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: MPV, n=7,3,22 | 0.00 (0.356) | 0.43 (0.808) | -0.11 (0.462)
  Day 113: MPV, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 113: MPV, n=7,3,19 | -0.04 (0.443) | 0.30 (0.781) | 0.03 (0.622)
  Day 155: MPV, n=6,3,17: number analyzed (Participants) | 6 | 3 | 17
  Day 155: MPV, n=6,3,17 | 0.17 (0.565) | 0.10 (0.872) | 0.01 (0.448)
  Day 197: MPV, n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: MPV, n=7,3,15 | -0.11 (0.385) | 0.10 (0.781) | 0.07 (0.580)

7. Primary Outcome: Change From Baseline in Hematology Parameters: Red Blood Cell (RBC) Count, Reticulocyte Count
Description: Blood samples were collected to analyze the hematology parameters: RBC count and reticulocyte count. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Tera cells per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Tera cells per liter
  Day 15: RBC count, n=8,3,23 | -0.05 (0.321) | 0.07 (0.208) | -0.01 (0.205)
  Day 29: RBC count, n=8,3,23 | -0.03 (0.225) | -0.07 (0.404) | -0.11 (0.275)
  Day 43: RBC count, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: RBC count, n=8,3,22 | -0.03 (0.238) | -0.07 (0.321) | -0.22 (0.331)
  Day 57: RBC count, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: RBC count, n=6,3,22 | -0.07 (0.288) | -0.10 (0.361) | -0.42 (0.464)
  Day 71: RBC count, n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: RBC count, n=8,3,20 | -0.13 (0.396) | -0.23 (0.208) | -0.66 (0.406)
  Day 85: RBC count, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: RBC count, n=7,3,22 | -0.10 (0.311) | -0.33 (0.208) | -0.68 (0.343)
  Day 113: RBC count, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: RBC count, n=7,3,20 | -0.13 (0.350) | -0.40 (0.265) | -0.68 (0.361)
  Day 155: RBC count, n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: RBC count, n=7,3,17 | -0.17 (0.330) | -0.37 (0.252) | -0.47 (0.264)
  Day 197: RBC count, n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: RBC count, n=7,3,15 | -0.04 (0.282) | -0.23 (0.058) | -0.15 (0.160)
  Day 15: Reticulocyte count, n=8,3,23 | 0.0109 (0.02401) | -0.0207 (0.02463) | -0.0160 (0.00964)
  Day 29: Reticulocyte count, n=8,3,23 | -0.0001 (0.00543) | -0.0169 (0.00911) | -0.0132 (0.01784)
  Day 43: Reticulocyte count, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Reticulocyte count, n=8,3,22 | -0.0032 (0.00554) | -0.0228 (0.02303) | -0.0109 (0.01699)
  Day 57: Reticulocyte count, n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: Reticulocyte count, n=6,3,22 | -0.0058 (0.00638) | -0.0091 (0.02177) | -0.0031 (0.01656)
  Day 71: Reticulocyte count, n=8,3,19: number analyzed (Participants) | 8 | 3 | 19
  Day 71: Reticulocyte count, n=8,3,19 | 0.0026 (0.01261) | -0.0125 (0.01878) | 0.0065 (0.01934)
  Day 85: Reticulocyte count, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: Reticulocyte count, n=7,3,22 | -0.0044 (0.00539) | -0.0209 (0.02471) | 0.0152 (0.02006)
  Day 113: Reticulocyte count, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: Reticulocyte count, n=7,3,20 | -0.0064 (0.01030) | 0.0012 (0.02944) | 0.0356 (0.02009)
  Day 155: Reticulocyte count, n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: Reticulocyte count, n=7,3,17 | 0.0006 (0.00623) | -0.0157 (0.02263) | 0.0158 (0.01340)
  Day 197: Reticulocyte count, n=7,3,16: number analyzed (Participants) | 7 | 3 | 16
  Day 197: Reticulocyte count, n=7,3,16 | 0.0003 (0.00550) | -0.0285 (0.03458) | 0.0017 (0.01003)

8. Primary Outcome: Change From Baseline in Hematology Parameter: Red Cell Distribution Width (RDW)
Description: Blood samples were collected to analyze the hematology parameter: RDW. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Percentage of width
  Day 15: n=8,3,23 | 0.04 (0.711) | -0.27 (1.050) | -0.26 (0.667)
  Day 29: n=8,3,23 | 0.24 (0.417) | -0.53 (1.704) | -0.47 (1.036)
  Day 43: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: n=8,3,22 | 0.25 (0.583) | -0.97 (1.650) | -0.47 (1.049)
  Day 57: n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: n=6,3,22 | -0.02 (0.578) | -0.83 (2.248) | 0.15 (1.331)
  Day 71: n=8,3,20: number analyzed (Participants) | 8 | 3 | 20
  Day 71: n=8,3,20 | 0.04 (0.725) | -0.23 (2.570) | 0.96 (2.040)
  Day 85: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: n=7,3,22 | -0.04 (0.663) | -0.20 (2.307) | 1.67 (1.792)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | 0.26 (0.748) | 0.73 (1.950) | 4.24 (2.737)
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | -0.09 (0.771) | 0.10 (1.916) | 2.86 (1.636)
  Day 197: n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: n=7,3,15 | -0.16 (1.286) | -0.57 (1.872) | 1.06 (1.375)

9. Primary Outcome: Change From Baseline in Reticulocyte Production Index
Description: Blood samples were collected to analyze the hematology parameter: Reticulocyte Production Index. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Reticulocyte Production Index (RPI) was calculated as 'Reticulocyte Production Index = Reticulocyte Count (percent [%]) multiply by (x) (hematocrit [%] divided by [/] 45) x 1/ reticulocyte maturation time'.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Unitless
  Day 15: n=8,3,23 | 0.2009 (0.49644) | -0.1787 (0.53867) | -0.2757 (0.20191)
  Day 29: n=8,3,23 | 0.0391 (0.09687) | -0.2397 (0.51850) | -0.2460 (0.35460)
  Day 43: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: n=8,3,22 | -0.0691 (0.11447) | -0.3437 (0.55192) | -0.2342 (0.34389)
  Day 57: n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: n=6,3,22 | -0.0763 (0.13476) | -0.2877 (0.48015) | -0.1933 (0.32326)
  Day 71: n=8,3,19: number analyzed (Participants) | 8 | 3 | 19
  Day 71: n=8,3,19 | 0.0154 (0.24560) | -0.4643 (0.13444) | -0.1344 (0.29111)
  Day 85: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: n=7,3,22 | -0.0831 (0.14906) | -0.4530 (0.48914) | -0.0112 (0.32736)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | -0.1006 (0.21168) | -0.2633 (0.29016) | 0.2826 (0.33003)
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | -0.0033 (0.24087) | -0.4720 (0.24857) | 0.1105 (0.28718)
  Day 197: n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: n=7,3,15 | -0.0296 (0.11222) | -0.5693 (0.43160) | 0.0087 (0.16995)

10. Primary Outcome: Change From Baseline Hematology Parameter: Reticulocytes
Description: Blood samples were collected to analyze the hematology parameter: reticulocytes. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Percentage of reticulocytes
  Day 15: n=8,3,23 | 0.0026 (0.00534) | -0.0053 (0.00551) | -0.0037 (0.00236)
  Day 29: n=8,3,23 | 0.0001 (0.00155) | -0.0040 (0.00265) | -0.0030 (0.00423)
  Day 43: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: n=8,3,22 | -0.0008 (0.00128) | -0.0057 (0.00611) | -0.0021 (0.00389)
  Day 57: n=6,3,22: number analyzed (Participants) | 6 | 3 | 22
  Day 57: n=6,3,22 | -0.0012 (0.00214) | -0.0023 (0.00551) | 0.0004 (0.00422)
  Day 71: n=8,3,19: number analyzed (Participants) | 8 | 3 | 19
  Day 71: n=8,3,19 | 0.0014 (0.00325) | -0.0027 (0.00551) | 0.0037 (0.00625)
  Day 85: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 85: n=7,3,22 | -0.0007 (0.00138) | -0.0043 (0.00651) | 0.0065 (0.00647)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | -0.0011 (0.00219) | 0.0013 (0.00702) | 0.0121 (0.00704)
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | 0.0006 (0.00162) | -0.0027 (0.00603) | 0.0054 (0.00405)
  Day 197: n=7,3,15: number analyzed (Participants) | 7 | 3 | 15
  Day 197: n=7,3,15 | 0.0001 (0.00157) | -0.0063 (0.00924) | 0.0005 (0.00233)

11. Primary Outcome: Number of Participants With Worst-Case Chemistry Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of clinical chemistry parameters. PCI ranges were low: <30 grams per liter (g/L) (albumin), high: >44.2 micromoles per liter (µmol/L) increase from Baseline (creatinine), low: <3 or high: >9 mmol/L (glucose), low: <3 or high: >5.5 mmol/L (potassium), and low: <130 or high: >150 mmol/L (sodium). Participants were counted in the worst case category that their value changes to (low, within range or no change, or high), unless there was no change in their category. Participants whose laboratory value category was unchanged (e.g. High to High), or whose value became within range, were recorded in the "To within Range or No Change" category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add up to 100%.
Time Frame: Up to Day 197
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Participants
  Albumin: To Low | 0 | 0 | 0
  Albumin: To within Range or No Change | 8 | 3 | 23
  Albumin: To High | 0 | 0 | 0
  Creatinine: To Low | 0 | 0 | 0
  Creatinine: To within Range or No Change | 8 | 3 | 23
  Creatinine: To High | 0 | 0 | 0
  Glucose: To Low | 0 | 0 | 1
  Glucose: To within Range or No Change | 8 | 2 | 19
  Glucose: To High | 0 | 1 | 3
  Potassium: To Low | 0 | 0 | 0
  Potassium: To within Range or No Change | 7 | 3 | 22
  Potassium: To High | 1 | 0 | 1
  Sodium: To Low | 0 | 0 | 0
  Sodium: To within Range or No Change | 8 | 3 | 23
  Sodium: To High | 0 | 0 | 0

12. Primary Outcome: Change From Baseline in Chemistry Parameter: Total Protein
Description: Blood samples were collected to analyze chemistry parameter: total protein. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Grams per liter
  Day 15: n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: n=7,2,23 | 1.0 (3.06) | 0.5 (4.95) | 0.4 (3.56)
  Day 29: n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: n=8,2,23 | -0.1 (3.14) | -1.0 (5.66) | 0.7 (2.86)
  Day 43: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: n=8,3,22 | -0.1 (2.36) | -0.3 (2.08) | -0.5 (3.52)
  Day 57: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: n=7,3,22 | 1.3 (2.29) | 1.3 (2.08) | -0.5 (3.65)
  Day 71: n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: n=8,3,21 | -0.1 (3.56) | 0.7 (1.15) | -1.1 (4.44)
  Day 85: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: n=8,3,22 | 0.3 (1.39) | 0.0 (2.00) | 0.3 (3.71)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | -0.9 (2.61) | 1.7 (0.58) | 0.2 (4.06)
  Day 155: n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 155: n=7,3,18 | -1.3 (1.25) | 3.0 (7.21) | -0.1 (4.59)
  Day 197: n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: n=7,3,19 | 2.3 (3.90) | 2.3 (3.51) | 1.5 (5.00)

13. Primary Outcome: Change From Baseline in Chemistry Parameters: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Lactate Dehydrogenase (LDH)
Description: Blood samples were collected to analyze chemistry parameters: ALP, ALT, AST and LDH. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
International units per liter
  Day 15: ALP, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: ALP, n=7,2,23 | -1.3 (10.53) | -1.0 (4.24) | 0.6 (5.67)
  Day 29: ALP, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: ALP, n=8,2,23 | -2.3 (7.89) | 4.5 (6.36) | -1.1 (10.94)
  Day 43: ALP, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: ALP, n=8,3,22 | -4.4 (12.36) | 0.7 (7.51) | -1.1 (9.00)
  Day 57: ALP, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: ALP, n=7,3,22 | -5.0 (13.23) | 3.3 (9.07) | 1.0 (7.55)
  Day 71: ALP, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: ALP, n=8,3,21 | -3.5 (10.94) | 1.3 (1.53) | -3.0 (11.52)
  Day 85: ALP, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: ALP, n=8,3,22 | -2.4 (11.96) | -2.3 (4.93) | -3.0 (11.65)
  Day 113: ALP, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: ALP, n=7,3,20 | -1.3 (4.99) | -2.3 (4.93) | -6.3 (8.15)
  Day 155: ALP, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 155: ALP, n=7,3,19 | -8.4 (15.88) | -3.3 (5.69) | -5.4 (9.84)
  Day 197: ALP, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: ALP, n=7,3,19 | -3.6 (12.16) | -4.0 (6.93) | -2.1 (11.03)
  Day 15: ALT, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: ALT, n=7,2,23 | -0.4 (2.70) | 0.0 (1.41) | 1.6 (3.85)
  Day 29: ALT, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: ALT, n=8,2,23 | 0.6 (1.85) | -2.0 (2.83) | 3.3 (9.58)
  Day 43: ALT, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: ALT, n=8,3,22 | 1.3 (3.15) | 4.0 (6.08) | 3.1 (10.70)
  Day 57: ALT, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: ALT, n=7,3,22 | -1.6 (1.27) | 2.0 (4.58) | 3.7 (10.03)
  Day 71: ALT, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: ALT, n=8,3,21 | 0.3 (2.82) | 3.0 (6.24) | 0.0 (2.67)
  Day 85: ALT, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: ALT, n=8,3,22 | -1.5 (3.89) | -0.3 (2.52) | 0.4 (4.27)
  Day 113: ALT, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: ALT, n=7,3,20 | -1.4 (5.13) | 4.7 (8.14) | 0.2 (3.18)
  Day 155: ALT, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 155: ALT, n=7,3,18 | -2.6 (6.65) | 1.0 (1.00) | 0.9 (3.95)
  Day 197: ALT, n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 197: ALT, n=7,3,21 | 3.6 (3.87) | -0.3 (2.52) | 2.4 (4.69)
  Day 15: AST, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: AST, n=7,2,23 | -0.1 (1.77) | 0.5 (0.71) | 1.7 (5.11)
  Day 29: AST, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: AST, n=8,2,23 | 1.8 (7.11) | 1.0 (1.41) | 2.0 (5.42)
  Day 43: AST, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: AST, n=8,3,22 | 1.6 (6.74) | 2.0 (3.61) | 0.9 (4.14)
  Day 57: AST, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: AST, n=7,3,22 | -0.6 (2.82) | 2.3 (3.06) | 2.0 (5.34)
  Day 71: AST, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: AST, n=8,3,21 | 1.9 (5.00) | 3.3 (4.93) | -0.3 (1.98)
  Day 85: AST, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: AST, n=8,3,22 | -0.8 (4.37) | 0.3 (2.31) | -0.2 (2.20)
  Day 113: AST, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: AST, n=7,3,20 | -2.7 (4.39) | 1.3 (4.04) | -0.9 (2.50)
  Day 155: AST, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 155: AST, n=7,3,18 | -5.0 (7.70) | 2.3 (0.58) | -0.6 (2.66)
  Day 197: AST, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: AST, n=7,3,19 | 0.1 (4.91) | 2.7 (0.58) | 1.2 (3.32)
  Day 15: LDH, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: LDH, n=7,2,23 | 4.1 (28.54) | -3.5 (51.62) | 18.4 (32.34)
  Day 29: LDH, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: LDH, n=8,2,23 | -7.0 (14.95) | 11.0 (0.00) | 20.9 (22.90)
  Day 43: LDH, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: LDH, n=8,3,22 | 12.1 (11.54) | 2.7 (30.62) | 27.2 (34.69)
  Day 57: LDH, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: LDH, n=7,3,22 | -5.1 (19.36) | 15.3 (31.02) | 22.4 (23.71)
  Day 71: LDH, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: LDH, n=8,3,21 | 10.5 (29.62) | 13.3 (26.95) | 32.7 (29.90)
  Day 85: LDH, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: LDH, n=8,3,22 | -2.5 (26.26) | 3.0 (11.53) | 24.9 (28.66)
  Day 113: LDH, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: LDH, n=7,3,20 | -17.6 (17.89) | 6.3 (25.50) | 14.2 (26.43)
  Day 155: LDH, n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: LDH, n=7,3,17 | -20.4 (32.67) | 1.0 (16.00) | 13.4 (12.63)
  Day 197: LDH, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: LDH, n=7,3,19 | -10.9 (27.97) | 0.3 (20.60) | 16.1 (21.91)

14. Primary Outcome: Change From Baseline in Chemistry Parameters: Total Bilirubin, Direct Bilirubin
Description: Blood samples were collected to analyze chemistry parameters: total bilirubin and direct bilirubin. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Micromoles per liter
  Day 15: Total bilirubin, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: Total bilirubin, n=7,2,23 | 0.571 (2.2254) | 2.000 (2.8284) | -0.957 (1.8944)
  Day 29: Total bilirubin, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: Total bilirubin, n=8,2,23 | -1.000 (2.8284) | -3.000 (1.4142) | -0.087 (1.8565)
  Day 43: Total bilirubin, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Total bilirubin, n=8,3,22 | -1.500 (1.4142) | -2.000 (2.0000) | -0.364 (1.4653)
  Day 57: Total bilirubin, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: Total bilirubin, n=7,3,22 | -0.286 (1.3801) | -2.000 (0.0000) | -0.636 (2.0827)
  Day 71: Total bilirubin, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: Total bilirubin, n=8,3,21 | 0.250 (1.9821) | -1.333 (1.1547) | -0.095 (2.1425)
  Day 85: Total bilirubin, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: Total bilirubin, n=8,3,22 | 0.250 (2.7124) | -2.000 (0.0000) | -0.364 (1.8138)
  Day 113: Total bilirubin, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: Total bilirubin, n=7,3,20 | 0.000 (3.2660) | -1.333 (1.1547) | 0.100 (1.5183)
  Day 155: Total bilirubin, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 155: Total bilirubin, n=7,3,18 | -1.143 (3.0237) | -3.333 (1.1547) | -1.604 (2.4901)
  Day 197: Total bilirubin, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 197: Total bilirubin, n=7,3,20 | 0.571 (2.7603) | -4.000 (0.0000) | -1.416 (1.6976)
  Day 15: Direct bilirubin, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: Direct bilirubin, n=7,2,23 | 0.0 (0.00) | 0.0 (0.00) | -0.4 (1.59)
  Day 29: Direct bilirubin, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: Direct bilirubin, n=8,2,23 | -0.3 (0.71) | 0.0 (0.00) | 0.0 (1.21)
  Day 43: Direct bilirubin, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Direct bilirubin, n=8,3,22 | -0.3 (0.71) | 0.0 (0.00) | -0.2 (1.05)
  Day 57: Direct bilirubin, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: Direct bilirubin, n=7,3,22 | 0.0 (0.00) | 0.0 (0.00) | -0.4 (1.18)
  Day 71: Direct bilirubin, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: Direct bilirubin, n=8,3,21 | -0.3 (0.71) | 0.0 (0.00) | -0.1 (1.18)
  Day 85: Direct bilirubin, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: Direct bilirubin, n=8,3,22 | -0.3 (0.71) | 0.0 (0.00) | -0.2 (1.05)
  Day 113: Direct bilirubin, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: Direct bilirubin, n=7,3,20 | 0.0 (1.15) | -0.7 (1.15) | -0.3 (0.98)
  Day 155: Direct bilirubin, n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: Direct bilirubin, n=7,3,17 | -0.3 (0.76) | 0.0 (0.00) | -0.2 (0.97)
  Day 197: Direct bilirubin, n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 197: Direct bilirubin, n=7,3,17 | 0.0 (0.00) | 0.0 (0.00) | -0.1 (1.11)

15. Primary Outcome: Change From Baseline in Chemistry Parameters: Cholesterol, Direct High-density Lipoprotein (HDL) Cholesterol, Low-density Lipoprotein (LDL) Cholesterol, Triglycerides
Description: Blood samples were collected to analyze chemistry parameters: cholesterol, direct HDL cholesterol, LDL cholesterol and triglycerides. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose) and Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 22
Millimoles per liter
  Cholesterol: n=8,3,22 | -0.125 (0.7474) | 0.067 (0.1258) | 0.450 (0.5780)
  Direct HDL Cholesterol: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Direct HDL Cholesterol: n=7,3,22 | -0.093 (0.1718) | -0.033 (0.0289) | -0.036 (0.2989)
  LDL Cholesterol: n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  LDL Cholesterol: n=7,3,21 | -0.091 (0.7376) | 0.110 (0.1200) | 0.274 (0.5011)
  Triglycerides: n=8,3,22 | 0.025 (0.3427) | -0.020 (0.0800) | 0.535 (0.8036)

16. Primary Outcome: Change From Baseline in Chemistry Parameter: Corrected Calcium, Urea
Description: Blood samples were collected to analyze chemistry parameters: corrected calcium and urea. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Millimoles per liter
  Day 15: Corrected calcium, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: Corrected calcium, n=7,2,23 | 0.011 (0.0540) | -0.020 (0.0566) | -0.013 (0.0725)
  Day 29: Corrected calcium, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: Corrected calcium, n=8,2,23 | -0.035 (0.0563) | -0.070 (0.0424) | -0.036 (0.0809)
  Day 43: Corrected calcium, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Corrected calcium, n=8,3,22 | -0.003 (0.0483) | -0.060 (0.0200) | -0.061 (0.0737)
  Day 57: Corrected calcium, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: Corrected calcium, n=7,3,22 | -0.003 (0.0509) | -0.060 (0.0721) | -0.069 (0.0827)
  Day 71: Corrected calcium, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: Corrected calcium, n=8,3,21 | -0.023 (0.0362) | -0.020 (0.0000) | -0.066 (0.0705)
  Day 85: Corrected calcium, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: Corrected calcium, n=8,3,22 | -0.043 (0.0599) | -0.027 (0.0808) | -0.049 (0.0689)
  Day 113: Corrected calcium, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: Corrected calcium, n=7,3,20 | -0.026 (0.0746) | 0.000 (0.0346) | -0.035 (0.0550)
  Day 155: Corrected calcium, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 155: Corrected calcium, n=7,3,18 | -0.037 (0.0678) | 0.000 (0.0346) | -0.034 (0.0508)
  Day 197: Corrected calcium, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: Corrected calcium, n=7,3,19 | 0.014 (0.0862) | -0.020 (0.0600) | -0.020 (0.0629)
  Day 15: Urea, n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: Urea, n=7,2,23 | 0.0714 (1.13389) | -2.0000 (0.00000) | 0.3043 (1.56481)
  Day 29: Urea, n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: Urea, n=8,2,23 | 0.0000 (1.13389) | -0.7500 (0.35355) | 0.3043 (1.67698)
  Day 43: Urea, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: Urea, n=8,3,22 | 0.4375 (1.08356) | -0.8333 (0.28868) | 0.3182 (1.34116)
  Day 57: Urea, n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: Urea, n=7,3,22 | -0.1429 (1.14434) | -0.8333 (0.76376) | 0.5682 (1.30289)
  Day 71: Urea, n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: Urea, n=8,3,21 | -0.1875 (1.30760) | -0.5000 (0.50000) | 0.0952 (1.50515)
  Day 85: Urea, n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: Urea, n=8,3,22 | -0.1875 (1.25178) | -0.1667 (0.76376) | 0.4091 (1.40269)
  Day 113: Urea, n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: Urea, n=7,3,20 | 0.2857 (1.70434) | -0.8333 (0.28868) | 0.4000 (1.47434)
  Day 155: Urea, n=7,3,18: number analyzed (Participants) | 7 | 3 | 18
  Day 155: Urea, n=7,3,18 | 0.2857 (1.75255) | -0.8333 (1.15470) | 0.0912 (1.52540)
  Day 197: Urea, n=7,3,19: number analyzed (Participants) | 7 | 3 | 19
  Day 197: Urea, n=7,3,19 | -0.0714 (2.11007) | -1.0000 (0.50000) | 0.1510 (1.76450)

17. Primary Outcome: Change From Baseline in Chemistry Parameter: Estimated Glomerular Filtration Rate
Description: Blood samples were collected to analyze chemistry parameter: estimated glomerular filtration rate. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliliter/minute/1.73 square meter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Milliliter/minute/1.73 square meter
  Day 15: n=7,2,23: number analyzed (Participants) | 7 | 2 | 23
  Day 15: n=7,2,23 | -6.4180 (10.28099) | 1.7630 (1.28693) | -0.7528 (9.25789)
  Day 29: n=8,2,23: number analyzed (Participants) | 8 | 2 | 23
  Day 29: n=8,2,23 | -4.3085 (8.34077) | -2.7765 (9.78424) | -1.5543 (9.55847)
  Day 43: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 43: n=8,3,22 | -0.4780 (9.34592) | -4.3223 (3.88914) | -3.4266 (6.99189)
  Day 57: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: n=7,3,22 | 1.3446 (7.12100) | 2.6893 (5.61068) | -5.1256 (7.41957)
  Day 71: n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: n=8,3,21 | -0.4405 (12.50899) | -0.9993 (5.98467) | -2.5432 (7.12712)
  Day 85: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: n=8,3,22 | -1.0010 (8.15284) | -7.1513 (6.77426) | -5.1038 (8.90164)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | -2.7351 (12.23546) | -0.2900 (6.19990) | -8.5267 (7.71222)
  Day 155: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 155: n=7,3,20 | -0.9239 (13.25672) | -3.9510 (5.74000) | -4.2795 (9.19612)
  Day 197: n=7,3,21: number analyzed (Participants) | 7 | 3 | 21
  Day 197: n=7,3,21 | -4.2733 (15.36640) | -7.7100 (8.47159) | -2.7185 (8.91665)

18. Primary Outcome: Number of Participants With Emergent Worst Case Urinalysis Results by Dipstick
Description: Urine samples were collected for the assessment of potential of hydrogen, specific gravity, glucose, ketones, occult blood and protein by dipstick method. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters: potential of hydrogen, specific gravity, glucose, ketones, occult blood and protein were categorized as 'any increase from Baseline', which imply any increase in their concentrations in the urine sample. Only participants with emergent worst case any increase from Baseline values are presented.
Time Frame: Up to Day 197
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Participants
  Potential of hydrogen, Any increase | 0 | 0 | 0
  Specific gravity, Any increase | 0 | 0 | 3
  Glucose, Any increase | 0 | 0 | 0
  Ketones, Any increase | 1 | 0 | 4
  Occult blood, Any increase | 2 | 0 | 3
  Protein, Any increase | 1 | 0 | 4

19. Primary Outcome: Number of Participants With Vital Signs Relative to Change From Baseline by Potential Clinical Importance (PCI) Criteria
Description: Systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR) were measured in a seated or semi-supine position after 5 minutes of rest using a completely automated device. PCI ranges were: SBP (increase or decrease from Baseline of >=40 millimeter of mercury [mmHg]), DBP (increase or decrease from Baseline of >=20 mmHg), and HR (increase or decrease from Baseline of >=30 beats per minute). Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment.
Time Frame: Baseline (Day 1: Pre-dose) and up to Day 197
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Participants
  DBP: Decrease >=20 | 2 | 0 | 2
  DBP: Increase >=20 | 0 | 0 | 1
  SBP: Decrease >=40 | 0 | 0 | 0
  SBP: Increase >=40 | 0 | 0 | 2
  HR: Decrease >=30 | 0 | 0 | 0
  HR: Increase >=30 | 1 | 0 | 2

20. Primary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured in a seated or semi-supine position after 5 minutes of rest. Baseline was defined as the pre-dose Day 1 assessment, unless unavailable, in which case it was the latest pre-dose assessment. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1: Pre-dose), Days 15, 29, 43, 57, 71, 85, 113, 155 and 197
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Degrees Celsius
  Day 15: n=8,3,23 | 0.037 (0.4689) | 0.400 (0.4359) | 0.117 (0.3833)
  Day 29: n=8,3,23 | 0.037 (0.3889) | 0.467 (0.6807) | 0.130 (0.3470)
  Day 43: n=8,3,23 | 0.012 (0.4121) | 0.033 (0.4163) | 0.039 (0.4197)
  Day 57: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: n=7,3,22 | 0.100 (0.2449) | 0.133 (0.3215) | 0.177 (0.4253)
  Day 71: n=8,3,21: number analyzed (Participants) | 8 | 3 | 21
  Day 71: n=8,3,21 | -0.112 (0.5303) | 0.267 (0.5132) | 0.186 (0.4328)
  Day 85: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: n=8,3,22 | 0.012 (0.3563) | 0.467 (0.5859) | -0.023 (0.3854)
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | -0.257 (0.3505) | 0.400 (0.6245) | 0.100 (0.4952)
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | -0.257 (0.3409) | 0.167 (0.5033) | 0.118 (0.6054)
  Day 197: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 197: n=7,3,17 | -0.143 (0.4860) | 0.267 (0.4933) | 0.212 (0.5122)

21. Primary Outcome: Number of Participants With Worst-case Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT intervals. Abnormal findings were categorized as clinically significant and not clinically significant. Clinically significant abnormal findings were those which were not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline abnormal ECG findings have been presented.
Time Frame: Up to Day 57
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 7 | 3 | 23
Participants
  Abnormal- not clinically significant | 3 | 2 | 10
  Abnormal- clinically significant | 0 | 0 | 1

22. Secondary Outcome: Plasma Concentrations of GSK2330811
Description: Blood samples were collected at the indicated time points for pharmacokinetic analysis of GSK2330811. Pharmacokinetic (PK) Population was defined as participants in the 'Safety' population who received an active dose and for whom a PK sample was obtained and analyzed.
Time Frame: Days 1, 15, 29, 57, 85, 113, 155 and 197
Population: PK Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 3 | 24
Nanogram per milliliter
  Day 1: n=3,24 | NA (NA) — Mean and standard deviation could not be calculated due to high proportion of non-quantifiable (NQ) values (more than [>] 30 percent [%] of values were imputed). | 0.0 (NA) — Mean and standard deviation could not be calculated due to high proportion of NQ values (>30% of values were imputed).
  Day 15: n=3,23: number analyzed (Participants) | 3 | 23
  Day 15: n=3,23 | 5510.7 (2455.19) | 16197.9 (6354.54)
  Day 29: n=3,23: number analyzed (Participants) | 3 | 23
  Day 29: n=3,23 | 7782.3 (1563.04) | 23407.0 (8830.49)
  Day 57: n=3,22: number analyzed (Participants) | 3 | 22
  Day 57: n=3,22 | 9868.7 (818.51) | 32645.7 (15225.01)
  Day 85: n=3,22: number analyzed (Participants) | 3 | 22
  Day 85: n=3,22 | 10993.0 (717.89) | 29254.4 (16911.55)
  Day 113: n=3,20: number analyzed (Participants) | 3 | 20
  Day 113: n=3,20 | 4123.0 (420.29) | 11087.1 (7661.76)
  Day 155: n=3,16: number analyzed (Participants) | 3 | 16
  Day 155: n=3,16 | 580.0 (408.47) | 2892.9 (4093.61)
  Day 197: n=3,17: number analyzed (Participants) | 3 | 17
  Day 197: n=3,17 | 114.0 (NA) — Mean and standard deviation could not be calculated due to high proportion of NQ values (>30% of values were imputed). | 729.2 (841.17)

23. Secondary Outcome: Concentration at the End of the Dosing Interval (Ctrough) of GSK2330811
Description: Blood samples were collected at the indicated time points for PK analysis of GSK2330811.
Time Frame: Days 1, 15, 29, 57, 85, 113, 155 and 197
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 3 | 22
Nanogram per milliliter | 10993.0 (717.89) | 29254.4 (16911.55)

24. Secondary Outcome: Apparent Clearance (CL/F) of GSK2330811
Description: Blood samples were collected at the indicated time points for PK analysis of GSK2330811. Data was analyzed by population pharmacokinetic methods using a non-linear mixed-effects modelling approach.
Time Frame: Days 1, 15, 29, 57, 85, 113, 155 and 197
Population: PK Population. Only those participants with data available at the specified time points were analyzed. CL/F was estimated based on population PK modelling on the combination of data of participants dosed with GSK2330811, as it was more appropriate due to limited dose range (100 mg and 300 mg).
Measure: Geometric Mean (95% Confidence Interval); unit: Liter per hour
Groups:
- GSK2330811 100 mg and GSK2330811 300 mg - Overall: Participants received subcutaneous injection of GSK2330811 100 mg and 300 mg on Day 1 and then every other week until the final dose on Day 71 (Week 10).
Arm/Group | GSK2330811 100 mg and GSK2330811 300 mg - Overall
Number analyzed (Participants) | 26
Liter per hour | 0.0147 [0.0132 to 0.0163]

25. Secondary Outcome: Apparent Volume of Distribution (Vss/F) of GSK2330811
Description: as for outcome 24
Time Frame: Days 1, 15, 29, 57, 85, 113, 155 and 197
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | GSK2330811 100 mg and GSK2330811 300 mg - Overall
Number analyzed (Participants) | 26
Liter | 3.25 [NA to NA] — The PK parameters were calculated by fitting a population PK model using the combined data of participants dosed with 100 mg and 300 mg of GSK2330811. Since a minimal model was utilized, the Vss/F value was fixed to a plasma physiological value obtained from the literature. Hence, a confidence interval cannot be provided for this parameter.

26. Secondary Outcome: Serum Level of Total Oncostatin M (OSM)
Description: Blood samples were collected at indicated timepoints for analysis of total OSM levels in serum. Per Protocol Population comprised of participants in the 'Safety' population who complied with the protocol.
Time Frame: Days 1, 15, 29, 57, 85, 113, 155 and 197
Population: Per Protocol Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Picogram per milliliter
  Day 1: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 1: n=8,3,22 | 22.110 [13.08 to 57.40] | 30.590 [6.19 to 38.71] | 27.455 [16.93 to 81.71]
  Day 15: n=8,3,23 | 28.175 [18.07 to 57.48] | 576.850 [417.28 to 696.18] | 721.020 [496.63 to 1482.91]
  Day 29: n=8,3,23 | 26.210 [12.84 to 48.82] | 499.540 [487.14 to 635.94] | 974.220 [398.94 to 2500.01]
  Day 57: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: n=7,3,22 | 34.700 [13.40 to 43.94] | 651.710 [554.93 to 971.25] | 1211.570 [636.83 to 2350.65]
  Day 85: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: n=8,3,22 | 17.275 [14.38 to 66.28] | 613.290 [555.09 to 1229.71] | 1357.645 [542.85 to 2500.01]
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | 23.350 [8.42 to 81.11] | 687.810 [419.04 to 935.76] | 1044.650 [186.06 to 2378.21]
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | 23.850 [13.13 to 43.07] | 206.900 [143.55 to 363.62] | 359.340 [58.13 to 1097.70]
  Day 197: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 197: n=7,3,17 | 28.800 [19.58 to 36.13] | 54.290 [40.96 to 137.88] | 142.830 [28.82 to 607.09]

27. Secondary Outcome: Serum Level of Free OSM
Description: Blood samples were collected at indicated timepoints for analysis of free OSM levels in serum.
Time Frame: Days 1, 15, 29, 57, 85, 113, 155 and 197
Population: as for outcome 26
Measure: Median (Full Range); unit: Picogram per milliliter
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Picogram per milliliter
  Day 1: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 1: n=8,3,22 | 19.72 [8.3 to 45.3] | 28.93 [4.5 to 36.8] | 20.74 [8.8 to 56.0]
  Day 15: n=8,3,23 | 23.85 [11.7 to 40.7] | 0.73 [0.73 to 0.73] | 0.73 [0.73 to 0.73]
  Day 29: n=8,3,23 | 19.35 [4.5 to 37.1] | 0.73 [0.73 to 0.73] | 0.73 [0.73 to 0.73]
  Day 57: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: n=7,3,22 | 27.62 [6.1 to 35.9] | 0.73 [0.73 to 0.73] | 0.73 [0.73 to 0.73]
  Day 85: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: n=8,3,22 | 12.37 [5.9 to 47.6] | 0.73 [0.73 to 0.73] | 0.73 [0.73 to 0.73]
  Day 113: n=7,3,20: number analyzed (Participants) | 7 | 3 | 20
  Day 113: n=7,3,20 | 16.78 [5.7 to 58.5] | 0.73 [0.73 to 0.73] | 0.73 [0.73 to 0.73]
  Day 155: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 155: n=7,3,17 | 14.54 [7.3 to 32.7] | 0.73 [0.73 to 0.73] | 0.73 [0.7 to 1.7]
  Day 197: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 197: n=7,3,17 | 18.43 [12.2 to 23.5] | 0.73 [0.73 to 0.73] | 0.73 [0.7 to 2.7]

28. Secondary Outcome: Number of Participants With Positive Anti-GSK2330811 Antibodies
Description: Serum samples were collected for the determination of anti-GSK2330811 antibodies (ADA) using a binding antibody detection assay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that were confirmed positive in the confirmation assay were reported as 'positive'.
Time Frame: Days 1, 15, 57, 85 and 197
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
Number analyzed (Participants) | 8 | 3 | 23
Participants
  Day 1: n=8,3,23 | 0 | 0 | 3
  Day 15: n=8,3,23 | 0 | 0 | 1
  Day 57: n=7,3,22: number analyzed (Participants) | 7 | 3 | 22
  Day 57: n=7,3,22 | 0 | 0 | 2
  Day 85: n=8,3,22: number analyzed (Participants) | 8 | 3 | 22
  Day 85: n=8,3,22 | 0 | 0 | 1
  Day 197: n=7,3,17: number analyzed (Participants) | 7 | 3 | 17
  Day 197: n=7,3,17 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-SAEs were collected up to Day 197. The protocol allowed for additional SAEs to be collected after Day 197; collected up to Day 603 post first dose
Description: Safety Population consisted of all randomized participants who have taken at least 1 dose of study treatment.
Arm/Group | Placebo | GSK2330811 100 mg | GSK2330811 300 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/3 | 2/24
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | GSK2330811 100 mg (N=3) | GSK2330811 300 mg (N=24)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | GSK2330811 100 mg (N=3) | GSK2330811 300 mg (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 2 (6)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (4) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 6 (6)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 2 (4)
Reticulocyte percentage increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Actinic elastosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Lentigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03041025/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03041025/SAP_001.pdf